CLINICAL TRIAL: NCT06466395
Title: A Phase I Study of Hyper-CVAD In Combination With Venetoclax In Pediatric Patients With Relapsed or Refractory Acute Leukemias That Are of the Lymphoid Lineage Including Bi-Phenotypic or Undifferentiated Leukemias
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-1044; NCI-2024-05154 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-06-14; First posted 2024-06-20 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Refractory Acute Leukemia; Relapsed Acute Leukemia; Undifferentiated Leukemia; Bi-Phenotypic Leukemia
MeSH Terms: interventions — venetoclax; CVAD protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1a (Experimental): Participants enrolled in Phase 1a, the dose of venetoclax the participant receive will depend on when the participant joins this study. The first group of participants will receive the lowest dose level of venetoclax. Each new group will receive a higher dose of venetoclax than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of venetoclax is found.
  The study doctor will discuss with you the doses the participants will receive as part of hyper-CVAD based on standard of care.
  Interventions: Drug: Venetoclax; Drug: Hyper-CVAD
- Phase 1b (Experimental): Participants enrolled in Phase 1b, will receive venetoclax at the recommended dose that was found in Phase 1.
  The study doctor will discuss with you the doses the participants will receive as part of hyper-CVAD based on standard of care.
  Interventions: Drug: Venetoclax; Drug: Hyper-CVAD

INTERVENTIONS:
Drug: Venetoclax — Given by PO
  Other Names: ABT-199; GDC-0199
Drug: Hyper-CVAD — Given by IV

SUMMARY:
To find the recommended dose of hyper-CVAD in combination with venetoclax that can be given to participants with relapsed or refractory leukemia.

DETAILED DESCRIPTION:
Primary Objectives

* To determine the maximum tolerated dose (MTD) and the recommended Phase 2 dose (RP2D) of venetoclax in combination with hyper-CVAD in patients with relapsed or refractory acute leukemias that are of the lymphoid lineage including bi-phenotypic or undifferentiated leukemias.
* To characterize the safety and tolerability of hyper-CVAD in combination with venetoclax.

Secondary Objectives

* To determine the preliminary assessment of efficacy by overall response (OR), including complete remission (CR), CR with incomplete blood count recovery (CRi) and partial response (PR).
* Evaluate additional measures of clinical benefit including overall survival (OS), event-free survival (EFS), progression-free survival (PFS) minimal residual disease (MRD) rate, and duration of response (DOR).

Exploratory Objectives

. To evaluate the pharmacodynamics (PD) and biological effects of hyper-CVAD in combination with venetoclax through molecular and cellular markers that may be predictive of antitumor activity and/or resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed/refractory leukemias as defined as:

   1. Pediatric, adolescent, or young adult patients with relapsed or refractory acute leukemias that are of the lymphoid lineage including bi-phenotypic or undifferentiated leukemias as per NCCN v2.2021 and W.H.O. classification in relapse or primary refractory.
   2. Participants must have ≥5% blasts in the bone marrow as assessed by morphology. However, if an adequate bone marrow sample cannot be obtained, patients may be enrolled if there is unequivocal evidence of leukemia with ≥5% blasts in the peripheral blood.
2. Participants have adequate performance status (ECOG ≤2) for patients ≥16 years old, Lansky score >50 for patients <16 years old.
3. Participants must be ≥ 2 years old or less than or equal to 21 years of age at time of signing/or having proxy sign the informed consent to be enrolled on study.
4. Participants with asymptomatic CNS disease are eligible.
5. These conditions are allowed on study: conditions requiring chronic systemic glucocorticoid use, such as autoimmune disease, graft versus host disease (GVHD) (well controlled on a stable dose of steroid or alternative therapy) or severe asthma. Participants are also allowed up to 5 days of glucocorticoids as cytoreduction, the use of hydroxyurea and the usage of cytarabine up to 2gm/m2. This should also be discussed with PI.

   1. For participants on chronic glucocorticoid therapy: Participants should be on stable systemic steroid doses less than or equal to 11.6mg/m2 (20 mg max) of prednisone daily

      * During times of dexamethasone dosing (cycles 1,3,5 and 7): Hold chronic steroids on days dexamethasone is given then resume normally scheduled chronic steroid dosing the following day.
      * Participants on chronic steroids > 11.6mg/m2 (20 mg max) prednisone equivalent will be excluded from the study.
   2. The use of topical steroids for cutaneous graft-versus-host disease (GVHD) is allowed.
   3. Participants should be at least 2 weeks or 5 half-lives (whichever is longer) from prior therapy, other than hydroxyurea, glucocorticoids or low dose cytarabine (as mentioned above) to maintain blast count prior to initiation of study therapy.
6. Participants must have adequate organ function and laboratory results (obtained within 14 days of enrollment):

   6.1. Total serum bilirubin ≤1.5 x upper limit of normal (ULN). Participants with known Gilbert's syndrome may have a total bilirubin up to ≤3 x ULN.

   6.2. Adequate renal function (creatinine clearance >30mL/min) unless related to the disease.

   6.3. Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≤3 x ULN; ≤5 x ULN unless in case of suspected leukemic liver involvement Females of childbearing potential must have a negative serum or urine beta-human chorionic gonadotropin (beta-hcg) pregnancy test result within 14 days prior to the first dose of study drugs and must agree to use one of the following effective contraception methods during the study and for 3 months following the last dose of study drug.

   The effects of these investigational agents on the developing human fetus are unknown. For this reason and because chemotherapeutic and inhibiting agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. This includes all female patients, between the onset of menses (as early as 8 years of age) and 55 years unless the patient presents with an applicable exclusionary factor which may be one of the following:
   * Postmenopausal (no menses in greater than or equal to 12 consecutive months).
   * History of hysterectomy or bilateral salpingo-oophorectomy.
   * Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).
   * History of bilateral tubal ligation or another surgical sterilization procedure.

     * Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
7. Males need to inform the doctor right away if the partner becomes pregnant or suspects pregnancy. While in this study and for 30 days after the last treatment the patient should not donate sperm for the purposes of reproduction. He will need to use a condom while in this study and for 30 days after the last treatment.
8. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of all study drug administration. Participants must have had at least 30 days between prior hematopoietic stem cell transplant and first dose of study drug.
9. For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
10. Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. For participants with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
11. Ability to understand and the willingness to sign a written informed consent document.
12. Participants with CD19+ B-ALL need to have received CD19-directed therapy prior to being considered for enrollment on this study.

Exclusion Criteria:

1. Past or current history of a secondary or other primary tumor or a chronic myeloid leukemia (CML) blast crisis with exception of:

   * curatively treated non-melanomatous skin cancer,
   * other primary solid tumor treated with curative intent and no known active disease present, and no treatment administered during the last 2 years.
2. Presence of clinically significant uncontrolled CNS pathology such as epilepsy, paresis, aphasia, stroke, severe brain injuries, organic brain syndrome, or psychosis.

   Presence of the following are allowed: headaches, vomiting, nerve palsy.
3. Significant traumatic injury or major surgery (major surgery means opening of a body cavity, e.g., thoracotomy, laparotomy, laparoscopic organ resection, and major orthopedic procedures, e.g. joint replacement, open reduction and internal fixation) within 14 days of scheduled dosing day 1.
4. Participants with uncontrolled infections (viral, bacterial, or fungal) per PI's discretion. Infections controlled on concurrent anti-microbial agents are acceptable, and anti-microbial prophylaxis per institutional guidelines are acceptable.
5. Medical history of cardiovascular disease such as:

   Clinically significant cardiac disease defined as congestive heart failure (NYHA class III or IV), arrhythmia or conduction abnormality requiring medication, or cardiomyopathy. This will be reviewed during screening EKG/ECHO as well as prior documentation.
6. Females who are pregnant or lactating.
7. Participants may be excluded if they are currently enrolled in another ongoing clinical trial with investigational products.
8. Liver cirrhosis or other active severe liver disease or with suspected active alcohol abuse.
9. Participants who are unable or unwilling to comply with all study requirements for clinical visits, examinations, tests, and procedures.
10. If participant has not recovered from previous chemotherapy, surgery, radiation before the start of study drugs.
11. Other severe, uncontrolled acute or chronic medical or psychiatric condition or laboratory abnormality that in the opinion of the Investigator may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and/or would make the patient inappropriate for enrollment into this study.
12. Participants with active/uncontrolled HIV infection, AIDS, or currently taking contraindicated medications for HIV control
13. History of allergic reactions attributed to compounds of similar chemical or biologic composition to all agents used in study. Since each reaction can vary from mild pruritis to anaphylaxis, the reaction will be discussed with PI prior to excluding participant.

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: David McCall, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org